CLINICAL TRIAL: NCT05518422
Title: Role of Endothelin-1 Modulating Insulin-stimulated Blood Flow and Sympathetic Nervous System Activity in Obesity
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jacqueline K Limberg, PhD, Assistant Professor, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2090413
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Insulin Resistance; Autonomic Dysfunction; Obesity
MeSH Terms: conditions — Insulin Resistance; Primary Dysautonomias; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral Bosentan (Experimental)
  Interventions: Drug: Hyperinsulinemic, euglycemic infusion

INTERVENTIONS:
Drug: Hyperinsulinemic, euglycemic infusion — 60 minute infusion

SUMMARY:
The aim of this project is to determine role for ET-1 in individuals with obesity.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years of age
* Male sex
* Obese (BMI ≥30 kg/m2)

Exclusion Criteria:

* Female sex
* Current smoking/Nicotine use
* Nerve/neurologic disease
* Cardiovascular, hepatic, renal, respiratory disease
* Blood pressure ≥140/90 mmHg
* Diabetes
* Vigorous exercise >3 times/week
* Communication barriers
* taking any medications known to affect metabolic, respiratory, cardiovascular, and/or autonomic

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Amount of muscle sympathetic nerve activity (MSNA) | Change from baseline at minute 60
  MSNA burst incidence (bursts/100 heart beats)
Amount of leg blood flow | Change from baseline at minute 60
  Measured with Doppler ultrasound (mL/min)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline K Limberg, Ph.D., Principal Investigator — University of Missouri-Columbia

IPD SHARING:
Plan to Share IPD: Undecided